CLINICAL TRIAL: NCT05513066
Title: Prospective, Observational and Bicentric Study of the Management of Arterial Hypotension During Planned Caesarean Section. Practice Comparison Between a Referral Center Using According to Service Protocol, an Intravenous Ephedrine/Phenylephrine Mixture at the PSE Versus Another Referral Center Using According to Service Protocol Intravenous Baby Noradrenaline
Brief Title: Management Arterial Hypotension During Planned Caesarean Section, Intravenous Ephedrine/Phenylephrine Mixture Versus Intravenous Baby Noradrenaline
Acronym: ARTEMIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: 2022 BONNIN ARTEMIS
Record Dates: First submitted 2022-08-19; First posted 2022-08-24 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-08

CONDITIONS: Hypotension
Keywords: cesarean; spinal anesthesia; hypotension; norepinephrine; ephedrine; phenylephrine; sympathetic block
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ephedrine/phenylephrine mixture: 10 mL of 0.75 mg/ml ephedrine and 10 mL of 37.5 μg/ml phenylephrine are mixed in a 20 mL syringe. The speed is generally started at 20 ml/h and then adapted according to blood pressure.
- baby noradrenaline: 20 mL of baby norepinephrine 10µg/mL is prepared in a 50 mL syringe. The speed is generally started at 30 ml/h and then adapted according to blood pressure.

SUMMARY:
Comparison of two practices of obstetrical services between the CHU of Clermont Ferrand and the HFME Lyon-Bron in the management of arterial hypotension during an elective cesarean section

DETAILED DESCRIPTION:
The investigators propose to carry out a bicentric strict observational prospective study between the maternity of the HFME of Lyon-Bron which uses the mixture ephedrine / noradrenaline with the PSE for many years in service protocol for the management of hypotension for cesarean section under perimedullary anesthesia and the CHU of Clermont-Ferrand which uses baby noradrenaline 10 mcg/mL PSE for this same indication according to an institutional protocol. Patients corresponding to the inclusion and non-inclusion criteria will be recruited by a physician investigator and will give their agreement of non-opposition after having received clear oral and written information about our study. The care will not be modified in any way compared to the usual practices of the service.

ELIGIBILITY:
Inclusion Criteria:

* elective caesarean
* ≥ 18 years old
* term ≥ 36 weeks amenorrhea

Exclusion Criteria:

* contraindication of local anesthetics
* contraindication of spinal anesthesia
* patient's refusal
* patient doesn't talk French
* patient not covered by the social security system

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients are included on their entry in the obstetrical operating room during an elective caesarean section if they meet the inclusion and exclusion criteria. The investigating doctor informs them of the terms of our purely observational research study before the intervention and asks them for their oral agreement.
  The study treatment administered depends on the protocol of the center in which they are included.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-09-02 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure | duration of the procedure up to one hour
  Time-weighted mean intraoperative systolic blood pressure below a threshold of 80mmHg, 90mmHg and 100mmHg. This measurement is commonly called TWA (time weighted average), corresponding to the area between the chosen PAS threshold and the curve of the measured PAS, divided by the total time of the measurements. Blood pressure will be measured by the Clearsight system, absolutely non-invasive continuous pulse wave contour monitoring.

SECONDARY OUTCOMES:
Clinical sign of hypotension | duration of the procedure up to one hour
  nausea, vomiting, faint
Foetal pH | at birth
  arterial and venous
boli of vasopressor | duration of the procedure up to one hour
  appeal to boli of ephedrine and/or phenylephrine and/or noradrenaline
boli of atropine | duration of the procedure up to one hour
  appeal to boli of atropine
crystalloids | duration of the procedure up to one hour
  volume of crystalloids infused
total diuresis | duration of the procedure up to one hour
intrathecal local anesthetics | duration of the procedure up to one hour
  amount of intrathecal local anesthetics injected

CONTACTS AND LOCATIONS:
Overall Officials: Martine BONNIN, Study Director — University Hospital, Clermont-Ferrand
Locations (2):
- France (2):
  - CHU clermont-ferrand, Clermont-Ferrand
  - Hospices Civils de Lyon, Lyon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee A, Ngan Kee WD, Gin T. A quantitative, systematic review of randomized controlled trials of ephedrine versus phenylephrine for the management of hypotension during spinal anesthesia for cesarean delivery. Anesth Analg. 2002 Apr;94(4):920-6, table of contents. doi: 10.1097/00000539-200204000-00028. PMID 11916798
- [Background] Lim G, Facco FL, Nathan N, Waters JH, Wong CA, Eltzschig HK. A Review of the Impact of Obstetric Anesthesia on Maternal and Neonatal Outcomes. Anesthesiology. 2018 Jul;129(1):192-215. doi: 10.1097/ALN.0000000000002182. PMID 29561267
- [Background] Vallejo MC, Attaallah AF, Elzamzamy OM, Cifarelli DT, Phelps AL, Hobbs GR, Shapiro RE, Ranganathan P. An open-label randomized controlled clinical trial for comparison of continuous phenylephrine versus norepinephrine infusion in prevention of spinal hypotension during cesarean delivery. Int J Obstet Anesth. 2017 Feb;29:18-25. doi: 10.1016/j.ijoa.2016.08.005. Epub 2016 Aug 28. PMID 27720613
- [Background] Yousif D, Bellos I, Penzlin AI, Hijazi MM, Illigens BM, Pinter A, Siepmann T. Autonomic Dysfunction in Preeclampsia: A Systematic Review. Front Neurol. 2019 Aug 6;10:816. doi: 10.3389/fneur.2019.00816. eCollection 2019. PMID 31447757
- [Background] Juri T, Suehiro K, Kimura A, Mukai A, Tanaka K, Yamada T, Mori T, Nishikawa K. Impact of non-invasive continuous blood pressure monitoring on maternal hypotension during cesarean delivery: a randomized-controlled study. J Anesth. 2018 Dec;32(6):822-830. doi: 10.1007/s00540-018-2560-2. Epub 2018 Sep 28. PMID 30267340
- [Background] Kinsella SM, Carvalho B, Dyer RA, Fernando R, McDonnell N, Mercier FJ, Palanisamy A, Sia ATH, Van de Velde M, Vercueil A; Consensus Statement Collaborators. International consensus statement on the management of hypotension with vasopressors during caesarean section under spinal anaesthesia. Anaesthesia. 2018 Jan;73(1):71-92. doi: 10.1111/anae.14080. Epub 2017 Nov 1. No abstract available. PMID 29090733
- [Background] Hollmen AI, Jouppila R, Koivisto M, Maatta L, Pihlajaniemi R, Puukka M, Rantakyla P. Neurologic activity of infants following anesthesia for cesarean section. Anesthesiology. 1978 May;48(5):350-6. doi: 10.1097/00000542-197805000-00009. PMID 646154
- [Background] Carvalho B, Dyer RA. Norepinephrine for Spinal Hypotension during Cesarean Delivery: Another Paradigm Shift? Anesthesiology. 2015 Apr;122(4):728-30. doi: 10.1097/ALN.0000000000000602. No abstract available. PMID 25654435
- [Background] Yu C, Gu J, Liao Z, Feng S. Prediction of spinal anesthesia-induced hypotension during elective cesarean section: a systematic review of prospective observational studies. Int J Obstet Anesth. 2021 Aug;47:103175. doi: 10.1016/j.ijoa.2021.103175. Epub 2021 May 1. PMID 34034957
- [Background] Ngan Kee WD, Lee SW, Ng FF, Tan PE, Khaw KS. Randomized double-blinded comparison of norepinephrine and phenylephrine for maintenance of blood pressure during spinal anesthesia for cesarean delivery. Anesthesiology. 2015 Apr;122(4):736-45. doi: 10.1097/ALN.0000000000000601. PMID 25635593
- [Background] Corke BC, Datta S, Ostheimer GW, Weiss JB, Alper MH. Spinal anaesthesia for Caesarean section. The influence of hypotension on neonatal outcome. Anaesthesia. 1982 Jun;37(6):658-62. doi: 10.1111/j.1365-2044.1982.tb01278.x. PMID 7091625
- [Background] Sklebar I, Bujas T, Habek D. SPINAL ANAESTHESIA-INDUCED HYPOTENSION IN OBSTETRICS: PREVENTION AND THERAPY. Acta Clin Croat. 2019 Jun;58(Suppl 1):90-95. doi: 10.20471/acc.2019.58.s1.13. PMID 31741565
- [Background] Singh PM, Singh NP, Reschke M, Ngan Kee WD, Palanisamy A, Monks DT. Vasopressor drugs for the prevention and treatment of hypotension during neuraxial anaesthesia for Caesarean delivery: a Bayesian network meta-analysis of fetal and maternal outcomes. Br J Anaesth. 2020 Mar;124(3):e95-e107. doi: 10.1016/j.bja.2019.09.045. Epub 2019 Dec 4. PMID 31810562